CLINICAL TRIAL: NCT03894384
Title: The Value of Serum Trefoil Factor Family 3 (TFF3) in Diagnosis of Gastric Cancer
Brief Title: The Value of TFF3 in Diagnosis of Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Melouk Ahmed, Director, Assiut University
Other Study IDs: TFF3 in gastric cancer
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-03

CONDITIONS: Gastric Cancer
Keywords: TFF3; PG1
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group:1: Gastric cancer patients
  Interventions: Diagnostic Test: Trefoil factor family 3 (TFF3),Pepsinogen 1(PG1)
- Group:2: Patients with benign gastric diseases
  Interventions: Diagnostic Test: Trefoil factor family 3 (TFF3),Pepsinogen 1(PG1)

INTERVENTIONS:
Diagnostic Test: Trefoil factor family 3 (TFF3),Pepsinogen 1(PG1) — Diagnostic Test: A) CBC . B) FBG. C)KFT. D) LFT. A)CBC: Complete blood count. B)FBG: Fasting blood glucose. C)KFT: Kidney function tests. D)LFT: Liver function tests.

SUMMARY:
Gastric cancer (GC), is a cancer developing from the inner lining of the stomach .The most common cause is infection by the bacterium Helicobacter pylori,which accounts for 60% of cases.

Human pepsinogens (HP) are proenzymes for pepsin; digestive enzymes produced by gastric chief cells, classified into two groups: pepsinogen I (PGI) and pepsinogen II (PGII), humen pepsinogens considered promising serological biomarkers for the screening of atrophic gastritis and gastric cancer.

The trefoil factor family (TFF) of peptides comprises small (12-22kDa) molecules that are secreted by the mammalian gastro-intestinal tract.Trefoil factor family 3 (TFF3) is a more stable non invasive biomarker of gastric cancer risk even in early gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer (GC), is a cancer developing from the inner lining of the stomach.Approximately half of the gastric cancer cases are diagnosed during advanced stages. One of the reasons for this is the invasiveness of esophagogastroduodenoscopy (EGD) screening examinations that leads to patients avoiding necessary tests .

The most common cause is infection by the bacterium Helicobacter pylori (H.pylori),which accounts for 60% of cases.

The development of tools for the early diagnosis of gastric cancer and precancerous lesions of gastric cancer is important for reducing mortality, increasing survival rates, and improving quality of life.

Endoscopy and biopsy are the reference standards for diagnosis and screening of gastric cancer, but their use is limited for population-wide screening due to their invasiveness.Subsequently, it is necessary to identify novel, simple, cost-effective and manipulable screening methods for gastric cancer.

Human pepsinogens (HP) are proenzymes for pepsin, a digestive enzymes produced by gastric chief cells,biochemically and immunochemically classified into two groups: pepsinogen I (PGI) and pepsinogen II (PGII), humen pepsinogens considered promising serological biomarkers for the screening of atrophic gastritis and gastric cancer,serum pepsinogen test provides a valuable method for detecting gastric cancer and atrophic gastritis.

The limitation of the pepsinogen test as a non invasive serologic biomarker screening method is that the optimal cut-off value could be affected by several factors, age, gender, and the test method itself.

The trefoil factor family (TFF) of peptides comprises small (12-22kDa) molecules that are secreted by the mammalian gastro-intestinal tract. TFFs constitute a family of three peptides (TFF1, TFF2, and TFF3) that are widely expressed in a tissue-specific manner in the gastro- intestinal tract. Trefoil factor family 3 (TFF3) is expressed in the goblet cells of the small and large intestines as well as the intestinal metaplasia in the stomach.

The trefoil factor family (TFF) plays a key role in the maintenance of mucosal integrity, and plays an impotant role in oncogenic transformation, growth, and metastatic extension of common human solid tumors, including gastric cancer.

SerumTFF3 showed good diagnostic power in both of H. pylori positive and H. pylori-negative gastric cancer and its serum levels were significantly higher in patients with advanced gastric cancer than that in patients with early gastric cancer.

H. pylori organisms live in gastric mucosa, and attach to epithelial cells of stomach .Because trefoil factor family 3 is not expressed in epithelial cells of the stomach and is only expressed in the intestinal goblet cells of the metaplasia of gastric cancer , serum trefoil factor family 3 levels are less influenced by H. pylori infection , eradication, aging, and sex ,therefore, serum trefoil factor family 3 is a more stable non invasive biomarker of gastric cancer risk even in early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Includes all patients presented by gastric cancer with clinical, radiological, laboratory diagnosis and pathological diagnosis.
* Individuals with benign diseases such as gastric polyps ,leiomyomas, gastric ulcers, atrophic gastritis and gastritis clinical, radiological, laboratory and pathological diagnosis.

Exclusion Criteria:

* - Previous upper gastrointestinal surgery, patients with gastric cancer that had been received chemotherapy, radiotherapy or surgical treatment.
* Patients simultaneously presented with a malignancy other than that of the stomach (Breast, pancreatic or colorectal).
* Pateints with severe systemic co-morbidities such as cardiopulmonary,hepatic and renal diseases

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted on 90 informed individuals (according to the guidelines of ethical committee of faculty of Medicine, Assiut University and South Egypt Cancer Institute).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of trefoil factor family 3 (TFF3) in serum of gastric cancer as non invasive marker | 2 day
  Measurement of TFF3 by enzyme linked immunosorbent assay (ELISA) in serum of gastric cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Heba Ahmed, MD, Principal Investigator — Assiut University; Ebtesam Farouk, MD, Study Chair — Assiut University; Abeer Ahmed, MD, Study Chair — Assiut University; Melouk Ahmed, Dr, Study Director — Assiut University
Locations (1):
- Melouk Ahmed Mahmoud, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi IJ. Endoscopic gastric cancer screening and surveillance in high-risk groups. Clin Endosc. 2014 Nov;47(6):497-503. doi: 10.5946/ce.2014.47.6.497. Epub 2014 Nov 30. PMID 25505714
- [Background] Lee JY, Park KS, Lee HG, Baek WK, Cho KB, Lee YJ, Lee YS, Ryu SW. Comparison of serum trefoil factor 3 with the pepsinogen test for the screening of diffuse-type gastric cancer. Clin Exp Med. 2017 Aug;17(3):403-410. doi: 10.1007/s10238-016-0426-1. Epub 2016 May 6. PMID 27154568
- [Background] Xiao P, Ling H, Lan G, Liu J, Hu H, Yang R. Trefoil factors: Gastrointestinal-specific proteins associated with gastric cancer. Clin Chim Acta. 2015 Oct 23;450:127-34. doi: 10.1016/j.cca.2015.08.004. Epub 2015 Aug 8. PMID 26265233